CLINICAL TRIAL: NCT06240975
Title: Comparative Effects of Theragun and Dry Needling on Neck Pain, Range of Motion and Disability Among Heavy Weightlifters
Brief Title: Theragun vs Dry Needling on Neck Pain, Range of Motion and Disability Among Heavy Weightlifters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0437
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Dry Needling; Neck Pain; Range of Motion; Weight Lifting
Keywords: Theragun; Dry Needling; Neck Pain; Range of Motion; Disability; Heavy weightlifters
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: randomized clinical trail
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theragun Technique (Other): Theragun is a handheld percussive therapy device that can be used for massage and muscle relaxation. Use the Theragun for a designated duration per session, such as 5-10 minutes for 6 weeks
  Interventions: Other: Theragun Technique
- Dry Needling Technique (Other): Dry needling is a technique in which a fine needle is used to penetrate the skin, subcutaneous tissues, and muscle without the use of an anesthetic. Hold each stretch for an adequate duration (typically 15-30 seconds) to allow for muscle relaxation
  Interventions: Other: Dry Needling Technique

INTERVENTIONS:
Other: Theragun Technique — Use the Theragun for a designated duration per session, such as 5-10 minutes for one session per week for 6 weeks
  Arms: Theragun Technique
Other: Dry Needling Technique — Dry needle deep (20 mm) TrP acupuncture of myofascial duration per session, such as 5-10 minutes for one session per week for 6 weeks
  Arms: Dry Needling Technique

SUMMARY:
The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive Theragun technique. Group B will receive Dry Needling technique.

DETAILED DESCRIPTION:
The objective of the study is to determine the Comparative effects of theragun and dry needling on neck pain, range of motion and disability among heavy weightlifters. The study is randomized and single-blinded. Ethical approval is taken from ethical committee of Riphah International University, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A & B through sealed envelope method by Non-probability Convenient random sampling technique. Subjects in Group A will receive Theragun technique. Group B will receive Dry Needling technique. Neck Disability index (NDI), Universal Goniometer, Numeric Pain Rating Scale (NPRS) will be used to assess at the baseline and after the completion of treatment at 6 weeks.

The data will be analyzed by SPSS, version 25. Statistical significance is P=0.05.

ELIGIBILITY:
Inclusion Criteria:

* •Male athlete,

  * 20 -35 years of age,
  * Weight lifting from 1 -2 years,
  * Cervical Flexion-Rotation Test positive

Exclusion Criteria:

* • Cerebrovascular diseases,

  * Migraine,
  * Cervicogenic Headache,
  * Musculoskeletal, cervical spondylosis, cervical spondylolisthesis,
  * Cervical post-operative,
  * Traumatic events in the past three months,
  * Presence of a physical or mental illness

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — healthy male athlete
Enrollment: 28 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Disability | pre and 6 weeks post interventional
  The Neck Disability Index (NDI) is commonly used for clinical and research assessment for chronic neck pain
Range of Motion | pre and 6 weeks post interventional
  A goniometer is an instrument that measures the available range of motion at a joint
Neck Pain | pre and 6 weeks post interventional
  Patient level of pain will be assessed using this Numerical Pain Rating Scale (NPRS)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Chand, DPT, Principal Investigator — Study Principal Investigator
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ariens GA, van Mechelen W, Bongers PM, Bouter LM, van der Wal G. Physical risk factors for neck pain. Scand J Work Environ Health. 2000 Feb;26(1):7-19. doi: 10.5271/sjweh.504. PMID 10744172
- [Background] Liu L, Huang QM, Liu QG, Ye G, Bo CZ, Chen MJ, Li P. Effectiveness of dry needling for myofascial trigger points associated with neck and shoulder pain: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):944-55. doi: 10.1016/j.apmr.2014.12.015. Epub 2015 Jan 7. PMID 25576642
- [Background] Pecos-Martin D, Montanez-Aguilera FJ, Gallego-Izquierdo T, Urraca-Gesto A, Gomez-Conesa A, Romero-Franco N, Plaza-Manzano G. Effectiveness of dry needling on the lower trapezius in patients with mechanical neck pain: a randomized controlled trial. Arch Phys Med Rehabil. 2015 May;96(5):775-81. doi: 10.1016/j.apmr.2014.12.016. Epub 2015 Jan 9. PMID 25582412
- [Background] Yang C, Huang X, Li Y, Sucharit W, Sirasaporn P, Eungpinichpong W. Acute Effects of Percussive Massage Therapy on Thoracolumbar Fascia Thickness and Ultrasound Echo Intensity in Healthy Male Individuals: A Randomized Controlled Trial. Int J Environ Res Public Health. 2023 Jan 7;20(2):1073. doi: 10.3390/ijerph20021073. PMID 36673829
- [Background] Hatefi M, Jaafarpour M, Khani A, Khajavikhan J, Kokhazade T. The Effect of Whole Body Massage on the Process and Physiological Outcome of Trauma ICU Patients: A Double-Blind Randomized Clinical Trial. J Clin Diagn Res. 2015 Jun;9(6):UC05-8. doi: 10.7860/JCDR/2015/12756.6096. Epub 2015 Jun 1. PMID 26266191
- [Background] Gattie E, Cleland JA, Snodgrass S. The Effectiveness of Trigger Point Dry Needling for Musculoskeletal Conditions by Physical Therapists: A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2017 Mar;47(3):133-149. doi: 10.2519/jospt.2017.7096. Epub 2017 Feb 3. PMID 28158962
- [Background] Sams L, Langdown BL, Simons J, Vseteckova J. The Effect Of Percussive Therapy On Musculoskeletal Performance And Experiences Of Pain: A Systematic Literature Review. Int J Sports Phys Ther. 2023 Apr 1;18(2):309-327. doi: 10.26603/001c.73795. eCollection 2023. PMID 37020441
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Fuentes-Gallardo I, Perez-Munoz M, Mayoral-Del-Moral O, Lluch-Girbes E, Prieto-Valiente L, Falla D. Effectiveness of dry needling for chronic nonspecific neck pain: a randomized, single-blinded, clinical trial. Pain. 2016 Sep;157(9):1905-1917. doi: 10.1097/j.pain.0000000000000591. PMID 27537209